CLINICAL TRIAL: NCT00552942
Title: Randomized Controlled Trial of Laparoscopic Gastric Bypass Plus Omentectomy Versus Laparoscopic Gastric Bypass Alone in Improving Diabetic Indices
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Legacy Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1234
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-11

CONDITIONS: Diabetes; Interleukins; Cytokines
Keywords: obesity; diabetes; cytokines
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): surgery plus omentectomy
  Interventions: Procedure: laparoscopic gastric bypass plus omentectomy
- 2 (No Intervention): standard gastric bypass

INTERVENTIONS:
Procedure: laparoscopic gastric bypass plus omentectomy
  Arms: 1

SUMMARY:
To see if removing the omentum in addition to a gastric bypass improves diabetes is better than just a gastric bypass.

ELIGIBILITY:
Inclusion Criteria:

* undergoing laparoscopic gastric bypass, >18 yo, understands english

Exclusion Criteria:

* previous lower pelvic surgery, self-pay patients, previous weight loss surgery,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
diabetic indices | 6 months

SECONDARY OUTCOMES:
interleukin and cytokine levels, weight loss | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hong, MD., MS.c, FRCSC, Principal Investigator — Oregon Weight Loss Surgery, LLC
Locations (1):
- Oregon Weight Loss Surgery LLC, Portland, Oregon, United States